CLINICAL TRIAL: NCT03487939
Title: Neoadjuvant FOLFOXIRI Chemotherapy in Resectable Liver Metastasis of Colorectal Cancer：an Open-label, Single-arm, Multicenter Phase II Study
Brief Title: Neoadjuvant FOLFOXIRI Chemotherapy in Resectable Liver Metastasis of Colorectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Medical University, China (Other)
Responsible Party: Principal Investigator, Jingdong Zhang, Director, China Medical University, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LGIOG-2017-03
Record Dates: First submitted 2018-03-24; First posted 2018-04-04 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Colorectal Neoplasms; Drug Therapy
MeSH Terms: conditions — Colorectal Neoplasms | interventions — FOLFOXIRI protocol; Irinotecan; Oxaliplatin; Fluorouracil

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FOLFOXIRI (Experimental): Patients received 4 cycles of neoadjuvant FOLFOXIRI chemotherapy before surgical resection.
  Interventions: Drug: FOLFOXIRI

INTERVENTIONS:
Drug: FOLFOXIRI — IRINOTECAN 150 mg/m^2 IV over 1-h, day 1 + OXALIPLATIN 85 mg/m^2 IV over 2-h, day 1 + L-LEUCOVORIN 200 mg/m^2 IV over 2-h, day 1 + 5-FLUOROURACIL 2800 mg/m^2 IV 48-h continuous infusion, starting on day 1 administered every two weeks for 4 cycles (2 months).
  Other Names: Irinotecan; Oxaliplatin; 5-Fluorouracil

SUMMARY:
To evaluate the efficacy and safety of neoadjuvant FOLFOXIRI chemotherapy (irinotecan, oxaliplatin and fluorouracil) in the patients with resectable liver metastasis of colorectal cancer

DETAILED DESCRIPTION:
For the patients Neoadjuvant FOLFOX chemotherapy is recommended for the resectable liver metastasis colorectal cancer. Neoadjuvant chemotherapy could suppress tumor, reduce metastasis, inhibit recurrence and improve long-term prognosis. Moreover, neoadjuvant chemotherapy could provide evidence about tumor response to drugs for the adjuvant chemotherapy. Furthermore, according to the biological behavior of tumors observed by neoadjuvant chemotherapy, unnecessarily excessive surgery could be avoided. However, some studies suggested that drug efficiency was consistent with resection rate. And FOLFOXIRI has been observed efficacy in the treatment of metastatic colorectal cancer with manageable toxicities. Therefore, we evaluate the efficacy and safety of neoadjuvant FOLFOXIRI chemotherapy in the patients with resectable liver metastasis of colorectal cancer to achieve higher resection rate and longer survival.

In this prospective study, 30 patients with resectable colorectal liver metastases were treated with neoadjuvant FOLFOXIRI chemotherapy. After 4 cycles of neoadjuvant chemotherapy, the liver metastases will be removed. If there are primary bowel lesions, they will be resected together. Safety profile was recorded based on NCI Common Terminology Criteria for Adverse Events version 4.0 (NCI-CTCAE v4.0). Objective response was evaluated by Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1). Before treatment and after 4 cycles of neoadjuvant chemotherapy, we will evaluate tumor metabolic response via FDG-PET and monitor the dynamic changes of peripheral blood ctDNA.

ELIGIBILITY:
Inclusion Criteria

* Age: 18-75years old
* Histologically confirmed colorectal cancer with liver metastasis (all patients should have the pathological report of colorectal cancer). The chances of hepatocellular carcinoma or metastasis from other primary lesions should be excluded.
* It was confirmed by imaging that the liver metastases and the primary intestinal lesions were all resectable.
* Radical resection of colorectal cancer after adjuvant chemotherapy complete 1 years later with liver metastases.
* There is at least one measurable objective tumor of the tumor (according to the 1.1 version of RECIST standard).
* Liver metastases can be excised by R0 and sufficient normal liver tissue can be retained
* ECOG status: 0～1
* Adequate bone marrow, hepatic and renal function as assessed by the following laboratory requirements conducted within 7 days of starting study treatment:

Neutrophil count≥1.5×10^9/L Platelet count≥90×10^9/L Hemoglobin≥90g/L Total bilirubin (TBI) ≤ 1.5 * ULN Alanine aminotransferase (ALT)≤2.5 * ULN Aspartate aminotransferase (AST)≤2.5 * ULN Alkaline phosphatase (ALP)≤2.5 * ULN

- Signed informed consent; able to comply with study and/or follow- up procedures

Exclusion Criteria:

* Hypersensitivity to fluorouracil, oxaliplatin or irinotecan.
* In addition to liver metastases, there are other parts of metastasis
* Cardiovascular disease that would preclude study treatment or follow-up; New York Heart Association class III or IV heart disease; Active ischemic heart disease; Myocardial infarction within the past 6 months; Symptomatic arrhythmia Uncontrolled hypertension. Unexplained syncope occurred within 3 months
* Gastric ulcers or duodenal ulcers for the treatment of resistance;
* 3 or 4 grade gastrointestinal bleeding / bleeding;
* Gastrointestinal perforation / fistula;
* Abdominal abscess;
* Infectious or inflammatory bowel disease
* HIV infection and/or active hepatitis B virus infection
* Pregnant or lactating women. Fertile patients must use effective contraception
* Any serious acute or chronic disease that can not be involved in the study or to influence the interpretation of the results of the study
* Other intervention clinical trials were combined at the same time.
* Nerve or mental abnormality affecting cognitive ability
* Other malignancy except effectively treated squamous cell or basal cell skin cancer,
* Other situations that the researchers think should be excluded.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2021-10-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
The ratio of tumor downstaging to stage 0 and stage I | 2 years
  Tumor downstaging from stage II or III to pathologic complete response (stage 0) and stage I

SECONDARY OUTCOMES:
Tumor regression grade (TRG) | 2 years
  The level of tumor regression under pathological examination
Disease free survival | 3 years
  Estimated from the date of surgery to the date of recurrence.
Overall survival time | 3 years
  Estimated from the date of enrollment to death from any cause.
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 3 years
  The grade of toxicity will be assessed using the NCI-CTCAE version 4.0.
ctDNA assessment and relation to clinical outcome | 3 years
  The relationship between ctDNA and survival will be evaluated.
SUVmax assessment and relation to clinical outcome | At the beginning of Cycle 1 and the end of Cycle 4 (each cycle is 14 days)
  Tumor metabolic response through FDG-PET examination before and after 4 cycles of neoadjuvant FOLFOXIRI chemotherapy
Quality of life (QLQ C30) | Every 2 weeks after the first treatment until 3 years
  Scores according to EORTC QLQ-C30 scoring manual

CONTACTS AND LOCATIONS:
Locations (1):
- Liaoning cancer hospital, Shenyang, Liaoning, China